CLINICAL TRIAL: NCT02248792
Title: Improvement in the Quality of Life of Patients With Severe Plaque Psoriasis Treated With Systemic Methotrexate in Fixed Doses of 10mg or 25mg Orally Once Weekly: a Prospective, Randomized, Double-blind, Parallel Group Study.
Brief Title: Quality of Life of Patients With Psoriasis Treated With Methotrexate: Prospective, Randomized, Double-blind, Parallel Group Study.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Narayana Medical College & Hospital (Other)
Responsible Party: Principal Investigator, C V Krishna, C V Krishna, Narayana Medical College & Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMCHDer
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Severe Plaque Type Psoriasis
MeSH Terms: interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Methotrexate 10mg orally once weekly
  Interventions: Drug: Methotrexate
- Group B (Active Comparator): Methotrexate 25mg orally once weekly
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate

SUMMARY:
Methotrexate (MTX) is considered the 'gold-standard' drug for the treatment of severe psoriasis. Health-related quality of life (HRQOL) is impaired in patients with psoriasis, more so if disease is severe.

ELIGIBILITY:
Inclusion Criteria:

Age range 18 to 65 years Both sexes Severe plaque-type psoriasis (BSA >10% or PASI >12) -

Exclusion Criteria:

Pregnancy Lactation Malignancy or immunosuppression including HIV Liver disease Renal disease Non compliant Psychiatric illness Hypersensitivity to methotrexate in the past

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in health related quality of life | 12 weeks

SECONDARY OUTCOMES:
comparison of improvement in health related quality of life between Group A and Group B | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: C V Krishna, MD, Principal Investigator — Narayana Medical college and hospital
Locations (1):
- Narayana Med College and Hospital, Nellore, Andhra Pradesh, India